CLINICAL TRIAL: NCT05237921
Title: Adherence to a Combined Exercise and Dietary Intervention in Patients With Gastrointestinal Cancer Undergoing Neo-adjuvant Therapy.
Brief Title: Adherence to Exercise and Dietary Intervention in Cancer Patients
Acronym: CEDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Beatriz Ângelo (Other)
Responsible Party: Principal Investigator, Sónia Velho, Nutricionist, Hospital Beatriz Ângelo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 178/18; 0261_B (Other: Hospital Beatriz Ângelo)
Record Dates: First submitted 2022-01-31; First posted 2022-02-14 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Adherence; Gastrointestinal Cancer
Keywords: Body composition; Wasting; Malnutrition
MeSH Terms: conditions — Gastrointestinal Neoplasms; Cachexia; Malnutrition | interventions — Diet Therapy; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Exercise and Dietary Intervention (Experimental): Behavioral Intervention
  Interventions: Behavioral: Combined Exercise and Dietary Intervention (CEDI)
- Control (Other): Standard Care
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Combined Exercise and Dietary Intervention (CEDI) — Intervention aimed at conveying a supervised combined moderate aerobic and resistance training, once a week with a duration of 40-60 minutes plus daily home exercise, personalized according to patients' age and functional status.
  Dietary intervention aimed at a one-on-one nutritional counseling. In the first visit a dietary plan is designed and one daily oral nutritional supplement (Forticare®, Nutricia) is given to meet the European Society of Parenteral and Enteral Nutrition (ESPEN) recommended intake.
  Arms: Combined Exercise and Dietary Intervention
Behavioral: Standard Care — Standard Care
  Arms: Control

SUMMARY:
Intervention programs in cancer patients have been proposed with the aim of improving outcome. Bearing in mind that compliance is a limiting factor to the benefit provided from exercise and diet, assessing adherence to these interventions is paramount before pursuing further studies. Therefore the purpose of this study was to study the adherence of gastrointestinal cancer patients to a Combined Exercise and Dietary Intervention (CEDI) during neo-adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with esophageal, gastric, pancreatic and rectal cancer
* Due to commence neo-adjuvant chemo/ radiotherapy (ChT)

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants that adhere to a Combined Exercise and Dietary Intervention (CEDI) | 8 weeks
  The aim of this study was to assess intervention adherence defined as the number of participants willing to engage in CEDI.

SECONDARY OUTCOMES:
Number of participants that meet estimated dietary intake and exercise goals | 8 weeks
  We will assess the number of participants able to achieve their estimated dietary goals, namely 25-30kcal/day and 1-1.5g protein day and at least attending to 50% of planed exercise sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Cravo, Study Director — Hospital da Luz
Locations (1):
- Hospital Beatriz Ângelo, Loures, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Study protocol with statistical analysis plan will be uploaded to trials.gov.
Supporting Information: Study Protocol, SAP

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT05237921/Prot_SAP_000.pdf